CLINICAL TRIAL: NCT04443777
Title: Analysis of Ergogenic Potential and Risks Associated With Acute and Chronic Use of Sulphonylureas on Physical Exercise
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Jocelito Bijoldo Martins, PhD student, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 5649/19
Record Dates: First submitted 2020-05-23; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Resistance Training; Sport Performance; Muscle Recovery; Hypoglycemic Agents; Randomized Controlled Trial
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, parallel-group clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulphonylurea Group (Active Comparator): Gliclazide 60 mg (Diamicron® MR) will be orally administered as matched capsules (same color, flavor, smell and size) 8 hours before the beginning of exercise session.
  Interventions: Other: Resistance Training
- Placebo Group (Placebo Comparator): Placebo (starch, sodium lauryl sulfate and Aerosil) will be orally administered as matched capsules (same color, flavor, smell and size) 8 hours before the beginning of exercise session.
  Interventions: Other: Resistance Training

INTERVENTIONS:
Other: Resistance Training — Both groups will perform the resistance training protocol that will consist of a warm-up on the bench press and leg press, both with workload at 50% of 1-RM. After a 2-minute rest, the resistance training session will be started. It will consist of 4 sets of bench press and leg press exercises at 65% of 1-RM with maximum repetitions until concentric failure, with the execution speed of 2x2. The bench press exercises will be followed by the leg press exercises with no interval between them. A 2-minute interval will allowed after each series of exercises.

SUMMARY:
This study have like aim to examine whether insulin secretagogues have a potential ergogenic effect leading to a better exercise performance and post-exercise recovery in healthy individuals after a resistance training session. METHODS: This is a randomized, double-blind, placebo-controlled, clinical trial. The sample will consist of 44 men. Subjects will be randomly allocated (block randomization, www.randomizer.org) to the following groups: placebo (PFG, n=22) and sulphonylurea (GFS, n=22). The study will consist of 3 visits 7 days apart. On visit 1 the participants will ask to sign an informed consent form and will carry out medical evaluation with anthropometric assessment. At that visit they will perform a one-repetition maximum test of the upper limbs by using the horizontal bench press and of the lower limbs by using the 45º leg press. On visit 2, they will perform a second round of similar 1-RM tests to determine workloads for the study session [sulphonylurea (gliclazide) vs. placebo]. The experimental exercise session will be held on visits 3. Gliclazide modified release 60 mg (Diamicron® MR) or placebo (starch, sodium lauryl sulfate and Aerosil) will be orally administered as matched capsules (same color, flavor, smell and size) 8 hours before the beginning of exercise session, double-blind. In the experimental session, first, warm-up on the bench press and leg press, both with workload at 50% of 1-RM will be carried out. After a 2-minute rest, the resistance training session will be started. It will consist of 4 sets of bench press and leg press exercises at 65% of 1-RM with maximum repetitions until concentric failure. The bench press exercises will be followed by the leg press exercises with no interval between them. A 2-minute interval will allowed after each series of exercises. Measurements for heart rate (HR) and Visual Analogue Scale (VAS) for Pain will be taken before, between each series of exercises and 24 and 48 hours after session. Venous blood samples will be obtained before, immediately after, 24 and 48 hours after, for determining serum levels of creatine kinase isoenzyme MM and lactate dehydrogenase. Capillary blood for glucose determination will be collected from the digital pulp using a glucometer before and immediately after. Resistance training volume will be calculated for each type of exercise as well as total training volume for each session as a product of exercise workload and number of series and repetitions.

DETAILED DESCRIPTION:
The use of performance-enhancing drugs is a major area of concern for high-performance athletes because it may lead to serious health problems. It is also quite concerning that these substances are also widely used without guidance among non-athletes for faster results and aesthetic reasons. Several substances used for doping in sports have well-established ergogenic and side effects. Studies have shown that insulin is used for its anabolic effects mostly among recreational and professional weightlifters and bodybuilders. Currently, insulin and its analogs are on the WADA list of prohibited substances for their anabolic effects mostly in muscle tissues and side effects. However, a class of drugs known as insulin secretagogues are used by some athletes to enhance performance. Few studies have examined the potential effects of insulin secretagogues, especially sulfonylureas, on exercise performance and post-exercise recovery among athletes as well as their potential side effects. Despite insufficient data supporting the use of insulin secretagogues as ergogenic supplement well as well its associated risks, these substances have been empirically used for both, acute and chronic effects among professional athletes and non-athletes. Thus, the present study have like aim to examine whether insulin secretagogues have a potential ergogenic effect leading to a better exercise performance and post-exercise recovery in healthy individuals after a resistance training session. METHODS: This is a randomized, double-blind, placebo-controlled, clinical trial. The sample will consist of 44 men, young adults, healthy and experienced in strength training and who meet the inclusion and exclusion criteria specified. The sample calculation was determined by a pilot study conducted with 10 subjects, with strength performance as the primary outcome, using drug (Gliclazide) or placebo, taking into account a statistical power of 95% and a significance level of 5%. For this purpose, the GPower 3.1was used. Subjects will be randomly allocated (block randomization, www.randomizer.org) to the following groups: placebo (PFG, n=22) and sulphonylurea (GFS, n=22). The study will consist of 3 visits 7 days apart. On visit 1 the participants will ask to sign an informed consent form and will carry out medical evaluation with anthropometric assessment. At that visit they will perform a one-repetition maximum test of the upper limbs by using the horizontal bench press and of the lower limbs by using the 45º leg press. On visit 2, they will perform a second round of similar 1-RM tests to determine workloads for the study sessions [sulphonylurea (gliclazide) vs. placebo]. The experimental exercise session will be held on visit 3. The participants will ask to follow a personalized food intake plan prescribed by a skilled provider in the 24 hours proceeding both sessions. Gliclazide modified release (MR) or placebo will be orally administered as matched capsules (same color, flavor, smell and size) 8 hours before the beginning of exercise session. Gliclazide 60 mg (Diamicron® MR) or placebo (starch, sodium lauryl sulfate and Aerosil) will administered double-blind. Upon arrival at the study site, the participants will consum a pre-workout snack. The experimental protocol will start 30 minutes later. First, warm-up on the bench press and leg press, both with workload at 50% of 1-RM wil be carried out. After a 2-minute rest, the resistance training session will be started. It will consist of 4 sets of bench press and leg press exercises at 65% of 1-RM with maximum repetitions until concentric failure, with the execution speed of 2x2. The bench press exercises will be followed by the leg press exercises with no interval between them. A 2-minute interval will allowed after each series of exercises. Measurements for heart rate (HR) and Visual Analogue Scale (VAS) for Pain will be taken before, between each series of exercises and 24 and 48 hours after session. Venous blood samples will be obtained before, immediately after, 24 and 48 hours after session for determining serum levels of creatine kinase isoenzyme MM and lactate dehydrogenase using a colorimetric enzymatic assay. Capillary blood for glucose determination will be collected from the digital pulp using a glucometer before and immediately after session. At the end of exercise session, a custom will be offered to prevent potential hypoglycemic events. Resistance training volume will be calculated for each type of exercise as well as total training volume for each session as a product of exercise workload and number of series and repetitions. The data will be present as means ± standard deviation (SD). Repeated measures ANOVA Two Way using Bonferroni post-hoc tests will be used for comparisons between the study drug and placebo over time. All data analyses will be carried out using SPSS 23.0 at a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* continuously resistance-trained for 2 years or more
* minimum frequency of 3 weekly sessions
* preceding 6 months

Exclusion Criteria:

* self-reported acute or chronic use of drugs including anabolic androgenic steroids, anti-inflammatory drugs, beta-blockers and exogenous insulin for the last 12 months
* alcohol intake within 72 hours of the study intervention
* injuries to bones and muscles preventing physical exercise
* non-adherence to dietary recommendations as instructed by the research team

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Resistance Training Performance | one week
  The performance of resistance training will be measured by the volume of training. This measure is obtained by the total load performed by the subject, measured in kilograms (Kg), being a product of the number of repetitions x the number of series and the load lifted by repetition (volume of training (Kg) = workload (Kg) x Repetition (nº) x Series (nº)). (18. Correa CS, Cadore EL, Martins JB, Silva ER, Pinto RS, Oliveira AR, Kruel LFM. The effects of ibuprofen on muscle performance, worload and plasma creatine kinase during strength training session. Medicina Sportiva. 2012;16(1):17-21).
Muscle Recovery Marker 1 | one week
  Serum levels of creatine kinase isoenzyme MM (CK-MM)
Muscle Recovery Marker 2 | one week
  Serum levels of lactate dehydrogenase (LDH)

SECONDARY OUTCOMES:
Subjective Perception Pain | one week
  Visual Analogue Scale (VAS) for Pain is a visual scale in which the subject reports how much pain the subject is feeling at the moment. This scale ranges from 0 to 10, where 0 means no pain and 10 means the greatest pain the subject has ever felt. It will be taken before, between each series of exercises and 24 and 48 hours after each session.The smaller the subjective sensation of pain, in this study, it will mean that recovery was faster and / or more effective.(16. Jensen M, Karoly P, Braver S. The measurement of clinical pain intensity: a comparision of six methods. Pain. 1986;27:117-26).
Blood Glucose Concentration | one week
  Capillary blood for blood glucose determination will be collected from the digital pulp using a glucometer (Free Style Optium) before and immediately after each session

CONTACTS AND LOCATIONS:
Locations (1):
- Fundação Universitária de Cardiologia/ Instituto de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martins JB, Zanella D, Nunes RB, Collado PS, Lehnen AM. Modified-release gliclazide acutely improves recovery but causes undesirable blood glucose decrease after a resistance exercise session in healthy adults: a pilot study for a randomized clinical trial. Arch Endocrinol Metab. 2024 Jul 30;68:e230381. doi: 10.20945/2359-4292-2023-0381. eCollection 2024. PMID 39420894